CLINICAL TRIAL: NCT00527527
Title: Chiropractic Dosage for Lumbar Stenosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University of Health Sciences (Other)
Collaborators: Foundation for Chiropractic Education and Research (FCER) (Other)
Responsible Party: Principal Investigator, Jerrilyn Cambron, DC, PhD, Researcher and Professor in the Dept of Research, National University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H0401
Record Dates: First submitted 2007-09-08; First posted 2007-09-11 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): 8 flexion distraction visits
  Interventions: Procedure: flexion distraction
- 2 (Active Comparator): 12 flexion distraction visits
  Interventions: Procedure: flexion distraction
- 3 (Active Comparator): 18 flexion distraction visits
  Interventions: Procedure: flexion distraction
- 4 (Placebo Comparator): 8 placebo control visits
  Interventions: Other: placebo control

INTERVENTIONS:
Procedure: flexion distraction — Chiropractic treatment using the flexion distraction apparatus
  Arms: 1; 2; 3
Other: placebo control — Placebo for comparison with flexion distraction treatment
  Arms: 4

SUMMARY:
This randomized clinical trial pilot study will investigate the efficacy of different amounts of total treatment dosage over six weeks in 60 volunteer subjects with lumbar spinal stenosis. Subjects will be evenly randomized into four groups of either flexion distraction (FD) care or a control: Group 1 with 8 total FD treatment visits, Group 2 with 12 total FD treatment visits, Group 3 with 18 total FD treatment visits, or Group 4 with 8 total placebo control visits. The study is designed: (1) To determine the feasibility of a larger scale study in terms of logistics, recruitment efforts, and sample size estimations and (2) To determine among the three treatment groups the change in perceived pain levels and general functional health status at the end of six weeks of treatment and at three months post care as follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 50 years old with lumbar spinal stenosis
* Impingement of the cord and/or exiting nerve roots evidenced on spine imaging studies
* Symptomatic with current pain in the back and/or one or both of the legs.
* Symptoms must have been present for at least six months with an insidious onset

Exclusion Criteria:

* Congenital stenosis or other spine deformities such as current spinal fractures, spinal infections, or tumors of the spine
* Prior lumbar spine surgery such as laminectomy, spinal fusion, or discectomy that lacks stability or occurred within the past 3 months.
* Currently pregnant or nursing
* Co-morbid conditions that may preclude a person from participating in active care (laying prone on a treatment table or completing exercises) and outcome measures (Treadmill Testing, completion of questionnaires), such as severe cardiopulmonary disorders (i.e.: severe coronary artery disease, recent myocardial infarction, or vascular claudication), neuromusculoskeletal disorders (i.e.: disabling hip or knee arthritis; trochanteric bursitis; piriformis syndrome; need for assisted ambulation), or brain disorders (i.e.: dementia or Alzheimer's Disease)
* Active conservative care such as physical therapy or chiropractic care for lumbar stenosis (excluding the use of oral medications or daily at-home exercises for general well-being)
* Cauda equina symptoms (i.e.: perianal numbness; loss of bowel and/or bladder control)
* Not fluent or literate in the English language. We will not be able to provide multiple translators within this pilot study
* Current or future litigation for low back or leg pain

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pain | 6 weeks; 3 and 6 months

SECONDARY OUTCOMES:
Functional health status | 6 weeks; 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jerrilyn Cambron, DC, PhD, Principal Investigator — National University of Health Sciences
Locations (1):
- National University of Health Sciences, Lombard, Illinois, United States